CLINICAL TRIAL: NCT01574313
Title: Effect of Stellate Ganglion Block on Meniere's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Yung-Song Lin, Chairman of department of Otolaryngology, Chi Mei Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGB09804-003; CMH09804-003 (Other Grant/Funding Number: Chi Mei Medical Center, Taiwan)
Record Dates: First submitted 2012-04-01; First posted 2012-04-10 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Vertigo; Meniere Disease
Keywords: stellate ganglion block.; Meniere's disease.; electrocochleography.; vertigo.; hearing impairment.
MeSH Terms: conditions — Vertigo; Meniere Disease; Hearing Loss | interventions — diphenidol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stellate ganglion block (Experimental): treated with SGB
  Interventions: Procedure: stellate ganglion block
- Oral medication (Active Comparator): treated with oral medications: 0.25mg of erispan@ (fludiazine) , 25mg cephadol@ (diphenidol), and 200mg kentons@ (tocopherol nicotinate).
  Interventions: Drug: 0.25mg, fludiazine; Drug: 25mg cephadol@ (diphenidol); Drug: 200mg kentons@ (tocopherol nicotinate).

INTERVENTIONS:
Procedure: stellate ganglion block — stellate ganglion block
  Arms: Stellate ganglion block
Drug: 0.25mg, fludiazine — 0.25mg of erispan@ (fludiazine), p.o. one dose only.
  Other Names: 0.25mg of erispan@
  Arms: Oral medication
Drug: 25mg cephadol@ (diphenidol) — 25mg cephadol@ (diphenidol) p.o. one dose only.
  Arms: Oral medication
Drug: 200mg kentons@ (tocopherol nicotinate). — 200mg kentons@ (tocopherol nicotinate) p.o. one dose only.
  Arms: Oral medication

SUMMARY:
Stellate ganglion block (SGB) has been the alternative treatment of Meniere's disease for years. However, objective evidence of the effect of SGB was still lack. The investigators conducted a randomized controlled study to examine the immediate effects of SGB in SP/AP of electrocochleography (ECoG).

DETAILED DESCRIPTION:
Ten patients were randomly assigned to receive stellate ganglion block. These ten patients made up the experimental group. Another ten patients in the control group were assigned to receiving one dosage of oral medications: 0.25mg of erispan@ (fludiazine) , 25mg cephadol@ (diphenidol), and 200mg kentons@ (tocopherol nicotinate).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with unilateral Meniere's disease, according to the criteria of the American Academy of Otolaryngology-Head and Neck Surgery, AAO-HNS (1995)

Exclusion Criteria:

* patients with coagulopathy,
* arrhythmia,
* myocardial ischemia,
* glaucoma,
* pregnant,
* chronic otitis media or externa, and
* past history of middle or inner ear surgery were excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
SP/AP of Electrocochleography | ECoG was reorded 2 hours after SGB
  SP/AP of ECoG was recorded 2 hours after SGB. to be compared with the SP/AP of ECoG recorded before treatment

SECONDARY OUTCOMES:
SP/AP recorded at 4 hours after SGB | 4 hours after SGB
  SP/AP recorded at 4 hours after SGB was compared with that of pretreatment with SGB
SP/AP recorded at 6 hours after SGB | 6 hours after SGB
  SP/AP recorded at 4 hours after SGB was compared with the SP/AP recorded before SGB
scores of verbal scale for vertigo recorded at 6 hours after SGB | 6 hours after SGB
  scores of verbal scale for vertigo recorded at 6 hours after SGB was compared to the scores recorded before SGB

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Song Lin, M.D., Principal Investigator — Chi Mei Medical Hospital
Locations (1):
- i Mei Medical Center Tainan, Taiwan, Taiwan, Tainan, Tainan, Taiwan